CLINICAL TRIAL: NCT02291237
Title: Study Title: A Phase 2/3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Effect of GS-6615 on Exercise Capacity in Subjects With Symptomatic Hypertrophic Cardiomyopathy
Brief Title: Effect of Eleclazine (GS-6615) on Exercise Capacity in Subjects With Symptomatic Hypertrophic Cardiomyopathy
Acronym: LIBERTY-HCM
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GS-US-361-1157; 2013-004429-97 (EudraCT Number)
Record Dates: First submitted 2014-11-11; First posted 2014-11-14 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2018-09-24 (Actual); Status verified 2018-02

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: hypertrophic cardiomyopathy; hcm; hocm; hypertrophic myocardiopathy; hypertrophic obstructive cardiomyopathies; cardiomyopathy; hypertrophic; familial hypertrophic cardiomyopathy; genetic heart disease; echocardiography; cardiopulmonary exercise testing; exercise Capacity; heart failure; angina; dyspnea; diastolic dysfunction; microvascular ischemia; late sodium current inhibitor; GS-6615; late INA
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathies; Hypertrophy; Cardiomyopathy, Hypertrophic, Familial; Heart Failure; Angina Pectoris; Dyspnea | interventions — eleclazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Eleclazine (Experimental): Eleclazine 30 mg single loading dose followed by 3 mg daily maintenance dose up until Week 12, then 6 mg daily maintenance dose from Week 12 at least Week 24, followed by eleclazine 6 mg in an open-label extension period.
  Interventions: Drug: Eleclazine
- Placebo (Experimental): Placebo to match eleclazine until at least Week 24, followed by active eleclazine 6 mg in an open-label extension period.
  Interventions: Drug: Eleclazine; Drug: Placebo

INTERVENTIONS:
Drug: Eleclazine — Tablet (s) administered orally once daily
  Other Names: GS-6615
Drug: Placebo — Placebo to match eleclazine administered orally once daily
  Arms: Placebo

SUMMARY:
The primary objective of this study was to evaluate the effect of eleclazine (GS-6615) on exercise capacity as measured by Peak oxygen uptake (VO2) achieved during cardiopulmonary exercise testing (CPET), in participants with symptomatic hypertrophic cardiomyopathy (HCM).

ELIGIBILITY:
Key Inclusion Criteria:

* Established diagnosis of hypertrophic cardiomyopathy defined by standard criteria as a maximal left ventricular wall thickness ≥ 15 mm at initial diagnosis
* Exertional symptoms including at least one of the following:

  * New York Heart Association (NYHA) Class ≥ II dyspnea
  * Canadian Cardiovascular Society (CCS) Class ≥ II angina
* Screening (baseline) peak VO2 < 80% of predicted for age, sex, and weight
* Ability to perform an upright treadmill cardiopulmonary exercise test (CPET)

Key Exclusion Criteria:

* Known aortic valve stenosis (moderate or severe)
* Known coronary artery disease
* Left ventricular systolic dysfunction (ejection fraction < 50%)
* Recent septal reduction procedure (ie, surgical myectomy or alcohol septal ablation) within six months prior to screening or such a procedure scheduled to occur during the study

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (46):
- United States (26):
  - Cedars-Sinai Heart Institute, Los Angeles, California
  - University of California Los Angeles, Los Angeles, California
  - Stanford University, Stanford, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Athens Regional Medical Center, Athens, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Brigham & Women's Hospital and Harvard Medical School, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - Tufts Medical Center, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University Medical Center/ New York Presbyterian, New York, New York
  - NYU School of Medicine Pediatrics, New York, New York
  - Duke Health Center at Southpoint, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - St. Luke's University Health Network, Bethlehem, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - St. Thomas Research Institute, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Texas Heart Institute, Houston, Texas
  - UT Southwestern Medical Center, Houston, Texas
  - University of Washington, Seattle, Washington
  - Marshfield Clinic Research Institute, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- The Alfred Hospital, Melbourne, Victoria, Australia
- Hôpital Européen Georges Pompidou, Paris, France
- Universitätsklinikum Hamburg Eppendorf, Hamburg, Germany
- Israel (4):
  - Ein Kerem-Hadassah Medical Organization, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (8):
  - Madonna del Soccorso Hospital, San Benedetto del Tronto, Ascoli Piceno
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero Universitaria Di Bologna, Bologna
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliera Monaldi, Naples
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Azienda Ospedaliera San Camillo Forlanini, Rome
- Netherlands (3):
  - Academisch Medisch Centrum Amsterdam, Amsterdam, North Holland
  - Erasmus MC, Rotterdam
  - University Medical Center Utrecht, Utrecht
- United Kingdom (2):
  - University Hospital of Wales, Cardiff, South Glamergon
  - Northern General Hospital, Sheffield, Yorkshire

REFERENCES:
- [Background] Olivotto I, Hellawell JL, Farzaneh-Far R, Blair C, Coppini R, Myers J, Belardinelli L, Maron MS. Novel Approach Targeting the Complex Pathophysiology of Hypertrophic Cardiomyopathy: The Impact of Late Sodium Current Inhibition on Exercise Capacity in Subjects with Symptomatic Hypertrophic Cardiomyopathy (LIBERTY-HCM) Trial. Circ Heart Fail. 2016 Mar;9(3):e002764. doi: 10.1161/CIRCHEARTFAILURE.115.002764. PMID 26915375

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Asia, Australia, Europe and North America. The first participant was screened on 05 February 2015. The last study visit occurred on 22 February 2017.
Pre-assignment Details: 264 participants were screened.
Groups:
- Eleclazine 30/3/6 mg: Single loading dose of eleclazine 30 mg (5 x 6 mg tablets) on Day 1, followed by 3 mg (1 x 3 mg tablet) daily maintenance dose until Week 12, then 6 mg (2 x 3 mg tablets) daily maintenance dose from Week 12 to at least Week 24
- Placebo: Placebo to match eleclazine administered orally for at least 24 weeks
Period: Overall Study
Arm/Group | Eleclazine 30/3/6 mg | Placebo
Started | 86 | 86
Completed | 0 | 0
Not Completed | 86 | 86
Not completed — Study Terminated by Sponsor | 72 | 67
Not completed — Adverse Event | 1 | 3
Not completed — Investigator's Discretion | 0 | 3
Not completed — Withdrew Consent | 11 | 11
Not completed — Lost to Follow-up | 0 | 2
Not completed — Subject Required Prohibited Medication | 2 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug
Groups:
- Placebo: Placebo to match eleclazine administered orally for up to at least 24 weeks
- Total: Total of all reporting groups
Arm/Group | Eleclazine 30/3/6 mg | Placebo | Total
Number analyzed (Participants) | 86 | 86 | 172
Age, Continuous [Mean (Standard Deviation); unit: years] | 46 (11.7) | 48 (10.3) | 47 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 36 | 73
  Male | 49 | 50 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 74 | 73 | 147
  Black or African American | 7 | 3 | 10
  Asian | 2 | 7 | 9
  Other | 2 | 1 | 3
  Not Permitted | 0 | 2 | 2
  American Indian or Alaska Native | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Or Latino | 11 | 9 | 20
  Not Hispanic Or Latino | 75 | 75 | 150
  Not Permitted | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 55 | 54 | 109
  Australia | 1 | 1 | 2
  France | 3 | 5 | 8
  Germany | 2 | 2 | 4
  Israel | 8 | 6 | 14
  Italy | 12 | 13 | 25
  Netherlands | 2 | 5 | 7
  United Kingdom | 3 | 0 | 3
Peak Oxygen Intake (VO2) [Mean (Standard Deviation); unit: mL/kg/min] — Population: Only 85 participants with available data from the placebo arm in safety analysis set were analyzed at baseline.
  mL/kg/min
    number analyzed (Participants) | 86 | 85 | 171
    (all) | 19.06 (4.853) | 19.88 (4.645) | 19.47 (4.755)

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Oxygen Uptake (VO2) Achieved During Cardiopulmonary Exercise Testing (CPET) From Baseline to Week 24
Time Frame: Baseline to Week 24
Population: Full Analysis Set: all randomized participants who received at least 1 dose of study drug. Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Eleclazine 30/3/6 mg | Placebo
Number analyzed (Participants) | 73 | 68
mL/kg/min | 0.15 (4.312) | 0.48 (4.143)
Statistical Analysis 1: Comparison: Eleclazine 30/3/6 mg vs Placebo; The analysis evaluated the change in Peak VO2 from baseline to Week 24 for the eleclazine group compared with that of the placebo group using analysis of covariance (ANCOVA) including terms for baseline Peak VO2, sex, and age (continuous); Test type: Superiority; p = 0.416, ANCOVA; P-value and Least Squares (LS) Means are from model with terms for sex, age (continuous), and treatment group and baseline peak VO2 as the covariate; LS Mean Difference(Eleclazine - Placebo) = -0.55, 95% CI 2-sided [-1.87 to 0.78]

2. Secondary Outcome: Change in Peak Oxygen Uptake (VO2) Achieved During Cardiopulmonary Exercise Testing (CPET) From Baseline to Week 12
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mL/kg/min
Arm/Group | Eleclazine 30/3/6 mg | Placebo
Number analyzed (Participants) | 83 | 78
mL/kg/min | 0.28 (4.028) | 0.57 (4.314)
Statistical Analysis 1: Comparison: Eleclazine 30/3/6 mg vs Placebo; The analysis evaluated the change in Peak VO2 from baseline to Week 12 for the eleclazine group compared with that of the placebo group using ANCOVA including terms for baseline Peak VO2, sex, and age (continuous); Test type: Superiority; p = 0.517, ANCOVA — P-value and LS Means are from model with terms for sex, age (continuous), and treatment group and baseline peak VO2 as the covariate; LS Mean Difference(Eleclazine - Placebo) = -0.42, 95% CI 2-sided [-1.68 to 0.85]

3. Secondary Outcome: Change in Minnesota Living With Heart Failure Questionnaire (MLHFQ) From Baseline to Week 24
Description: The MLHFQ is a 21-item quality of life (QoL) questionnaire that measures the effects of symptoms, functional limitations, and psychological distress on an individual. Each item is measured on a 6-point Likert scale (0 to 5) and is scored by summing the responses to all 21 questions. Scores range from 0 to 105, with lower scores indicating a better quality of life.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Eleclazine 30/3/6 mg | Placebo
Number analyzed (Participants) | 86 | 86
Score
  Baseline | 40.22 (25.544) | 38.80 (23.177)
  Change from Baseline at Week 24: number analyzed (Participants) | 74 | 73
  Change from Baseline at Week 24 | -4.05 (15.164) | -5.57 (14.345)
Statistical Analysis 1: Comparison: Eleclazine 30/3/6 mg vs Placebo; The analysis evaluated the change in MLHFQ from baseline to Week 24 for the eleclazine group compared with that of the placebo group using ANCOVA including terms for baseline treadmill exercise time, sex, and age (continuous); Test type: Superiority; p = 0.513, ANCOVA; P-value and LS Means are from model with terms for sex, age (continuous), and treatment group and baseline score as the covariate; LS Mean Difference(Eleclazine - Placebo) = 1.54, 95% CI 2-sided [-3.11 to 6.19]

4. Secondary Outcome: Change in Minnesota Living With Heart Failure Questionnaire (MLHFQ) From Baseline to Week 12
Description: as for outcome 3
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | Eleclazine 30/3/6 mg | Placebo
Number analyzed (Participants) | 86 | 86
Score
  Baseline | 40.22 (25.544) | 38.80 (23.177)
  Change at Week 12: number analyzed (Participants) | 85 | 80
  Change at Week 12 | -3.84 (15.654) | -3.40 (13.780)
Statistical Analysis 1: Comparison: Eleclazine 30/3/6 mg vs Placebo; The analysis evaluated the change in MLHFQ from baseline to Week 12 for the eleclazine group compared with that of the placebo group using ANCOVA including terms for baseline treadmill exercise time, sex, and age (continuous); Test type: Superiority; p = 0.964, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference(Eleclazine - Placebo) = 0.10, 95% CI 2-sided [-4.36 to 4.56]

5. Secondary Outcome: Change in Treadmill Exercise Time From Baseline to Week 24
Description: Treadmill exercise time is the time to peak exercise.
Time Frame: Baseline to Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Eleclazine 30/3/6 mg | Placebo
Number analyzed (Participants) | 86 | 86
min
  Baseline: number analyzed (Participants) | 86 | 84
  Baseline | 12.88 (4.641) | 13.60 (4.317)
  Change from Baseline at Week 24: number analyzed (Participants) | 73 | 68
  Change from Baseline at Week 24 | 0.27 (3.954) | 0.24 (3.208)
Statistical Analysis 1: Comparison: Eleclazine 30/3/6 mg vs Placebo; The analysis evaluated the change in treadmill exercise time from baseline to Week 24 for the eleclazine group compared with that of the placebo group using ANCOVA including terms for baseline treadmill exercise time, sex, and age (continuous); Test type: Superiority; p = 0.944, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference(Eleclazine - Placebo) = -0.04, 95% CI 2-sided [-1.18 to 1.10]

6. Secondary Outcome: Change in Treadmill Exercise Time From Baseline to Week 12
Description: Treadmill exercise time is the time to peak exercise.
Time Frame: Baseline to Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Eleclazine 30/3/6 mg | Placebo
Number analyzed (Participants) | 86 | 86
min
  Baseline: number analyzed (Participants) | 86 | 84
  Baseline | 12.88 (4.641) | 13.60 (4.317)
  Change from Baseline at Week 12: number analyzed (Participants) | 83 | 77
  Change from Baseline at Week 12 | 0.48 (3.295) | 0.38 (3.030)
Statistical Analysis 1: Comparison: Eleclazine 30/3/6 mg vs Placebo; The analysis evaluated the change in treadmill exercise time from baseline to Week 12 for the eleclazine group compared with that of the placebo group using ANCOVA including terms for baseline treadmill exercise time, sex, and age (continuous); Test type: Superiority; p = 0.993, ANCOVA; [statistical method as in outcome 3, analysis 1]; LS Mean Difference(Eleclazine - Placebo) = 0.00, 95% CI 2-sided [-0.96 to 0.97]

ADVERSE EVENTS:
Time Frame: Baseline up to the last dose date plus 30 days (maximum exposure: 668 days)
Description: Safety Analysis Set: all randomized participants who received at least 1 dose of study drug
Arm/Group | Eleclazine 30/3/6 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/86 | 0/86
Serious Adverse Events (participants affected / at risk) | 14/86 | 16/86
Other Adverse Events (participants affected / at risk) | 58/86 | 62/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eleclazine 30/3/6 mg (N=86) | Placebo (N=86)
ATRIAL FIBRILLATION (Cardiac disorders) | 2 | 1
ATRIAL FLUTTER (Cardiac disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE ACUTE (Cardiac disorders) | 1 | 0
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 2 | 0
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 1
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 3
HYPERTROPHIC CARDIOMYOPATHY (Congenital, familial and genetic disorders) | 0 | 1
CHEST PAIN (General disorders) | 2 | 2
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 1 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 1 | 0
CELLULITIS (Infections and infestations) | 0 | 1
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 1 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 2 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1
ENDOCARDITIS (Infections and infestations) | 1 | 0
ESCHERICHIA URINARY TRACT INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0
INFLUENZA (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
FOOT FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 1 | 0
SCAPULA FRACTURE (Injury, poisoning and procedural complications) | 1 | 0
CARDIAC INDEX DECREASED (Investigations) | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 1
SYNCOPE (Nervous system disorders) | 0 | 1
ANXIETY (Psychiatric disorders) | 0 | 1
SUICIDE ATTEMPT (Psychiatric disorders) | 0 | 1
CYSTITIS INTERSTITIAL (Renal and urinary disorders) | 0 | 1
URETEROLITHIASIS (Renal and urinary disorders) | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eleclazine 30/3/6 mg (N=86) | Placebo (N=86)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 6
PALPITATIONS (Cardiac disorders) | 9 | 11
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 2 | 5
NAUSEA (Gastrointestinal disorders) | 11 | 11
CHEST DISCOMFORT (General disorders) | 6 | 3
CHEST PAIN (General disorders) | 11 | 9
FATIGUE (General disorders) | 9 | 7
BRONCHITIS (Infections and infestations) | 1 | 5
INFLUENZA (Infections and infestations) | 3 | 5
NASOPHARYNGITIS (Infections and infestations) | 5 | 11
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 10
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 7
BACK PAIN (Musculoskeletal and connective tissue disorders) | 9 | 6
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 | 6
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 5
DIZZINESS (Nervous system disorders) | 12 | 14
HEADACHE (Nervous system disorders) | 11 | 11
HYPOAESTHESIA (Nervous system disorders) | 1 | 5
PRESYNCOPE (Nervous system disorders) | 5 | 8
ANXIETY (Psychiatric disorders) | 5 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 16 | 8

LIMITATIONS AND CAVEATS:
The totality of the data did not support continuation of the eleclazine development program. So, this study was terminated prior to the end of the double-blind phase, and therefore no participants entered the open-label extension (OLE) period.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (5):
  • Study Protocol: Original (2014-04-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT02291237/Prot_005.pdf
  • Study Protocol: Amendment 1 (2014-10-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT02291237/Prot_006.pdf
  • Study Protocol: Amendment 2 (2015-02-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT02291237/Prot_007.pdf
  • Study Protocol: Amendment 3 (2016-08-12): https://cdn.clinicaltrials.gov/large-docs/37/NCT02291237/Prot_008.pdf
  • Statistical Analysis Plan (2017-05-10): https://cdn.clinicaltrials.gov/large-docs/37/NCT02291237/SAP_009.pdf